CLINICAL TRIAL: NCT01545063
Title: Prospective Non-interventional Non-controlled Multicenter Observational Study to Evaluate the Quality of Care for Adult Patients on Home Parenteral Nutrition (HPN)
Brief Title: CAre of Patients With PArenteral Nutrition At Home
Acronym: CAPANAH
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Ziekenhuis Netwerk Antwerpen (ZNA) (Other); AZ Sint-Lucas Brugge (Other); Universiteit Antwerpen (Other); AZ Sint-Blasius Dendermonde (Unknown); Imelda Hospital, Bonheiden (Other); Ziekenhuis Oost-Limburg (Other); AZ Damiaan, Oostende (Unknown); H.-Hartziekenhuis Roeselare-Menen vzw (Unknown); Universitair Ziekenhuis Brussel (Other); University Hospital, Ghent (Other); Jessa Hospital (Other)
Responsible Party: Principal Investigator, Mira Dreesen, PhD student, PhD Student, KU Leuven
Other Study IDs: S54137
Record Dates: First submitted 2012-03-01; First posted 2012-03-06 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Crohn's Disease; Peritoneal Carcinomatosis With Intestinal Occlusion; Radiation Enteritis; Chronic Diarrhea; Intestinal Lymphomas
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research aims to give an overview of a number of aspects related to the quality of care for adult patients on home parenteral nutrition.

Concretely this study follows up different aspects on different moments in the care of the patient pathways:

* process indicators concerning indication, parenteral nutrition, training, team access roads and the succession of complications
* Outcome indicators
* the health-related quality of life
* discrepancies in medication use
* the role of the different health care providers

DETAILED DESCRIPTION:
Adult patients on HPN will be contacted by phone at three different time moments after their discharge to ask them about indicators, quality of life and discrepancies in medication use. After the follow-up, medical dossiers will be consulted to know which indicators are followed in practice.

The role of the different health care providers will be investigated by face-to-face interviews with different healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* Patients in Flanders who speak Dutch, are older then 18 years and are able to give an informed consent.

Exclusion Criteria:

* Patients who are younger then 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult HPN patients with peritoneal carcinomatosis with intestinal occlusion or with crohn's disease, radiation enteritis, chronic diarrhea, intestinal lymphomas.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Quality of life | 2 years
  Quality of life will be investigated with the HPN-QoL(r) or FACIT-G (r).
Number of catheter related infections | 2 years

CONTACTS AND LOCATIONS:
Locations (13):
- Belgium (13):
  - Antwerpen Middelheim, Antwerp
  - UZA Antwerpen Edegem, Antwerp
  - Imelda Ziekenhuizen Bonheide, Bonheiden
  - AZ Sint-Lucas, Bruges
  - University Centrum Brussel, Brussels
  - AZ Sint Blasius Dendermonde, Dendermonde
  - Ziekenhuis Oost Limburg, Genk
  - AZ Sint Lucas en Volkskliniek, Ghent
  - UZ Gent, Ghent
  - Hasselt Jessa Ziekenhuizen, Hasselt
  - Catholic University, Leuven
  - AZ Damiaan, Ostend
  - Heilig Hart vzw, Roeselare Menen

IPD SHARING:
Plan to Share IPD: No